CLINICAL TRIAL: NCT04716023
Title: Physiology and Structure of the Small Airways in Patients With Chronic Airflow Obstruction or COVID-19
Acronym: PASSPORT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 18IC4688
Record Dates: First submitted 2020-07-02; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Copd; COVID-19; Asthma; Small Airways Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; COVID-19; Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic Airflow obstruction / COVID-19: Patients with either chronic airflow obstruction of COVID-19

SUMMARY:
The purpose of this research project is to study small airways physiological function in patients with chronic obstructive lung disease or COVID-19 and explore the relationship with in-vivo microanatomical small airway structure as measured by OCT. Correlating endobronchial assessment with multiple breath nitrogen washout and impulse oscillometry will allow the characterisation of the relationship between small airway structural findings and these validated investigations. A small volume lung wash, endobronchial brushings and the collection of a limited number of endobronchial cryobiopsy samples will be performed to better understand the endobronchial environment of the small airways through inflammatory studies. Following the completion of any such work, residual samples will be stored in a "bio-bank" to enable the completion of future work. Understanding the relationship with symptom-based quality of life scoring questionnaires and a functional assessment of exercise capacity will help elucidate the clinical impact of in-vivo small airways findings.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16 or over
2. Scheduled for bronchoscopy as part of clinical care or research protocol
3. No bleeding diathesis or therapeutic anticoagulation
4. COPD:

   * FEV1/FVC ratio <70% or

Asthma:

* Diagnosed by standard clinical methods
* Post-bronchodilator FEV1 ≥60% predicted or COVID-19 infection or previous COVID-19 infection (confirmed as per local guidelines)

Exclusion Criteria:

1. Unable to provide informed consent
2. Exacerbation of obstructive airways disease or respiratory infection requiring systemic antibiotics or corticosteroids in the 6 weeks prior to enrolment unless suffering from COVID-19 infection and bronchoscopy is required for clinical reasons
3. Contra-indications to performing lung function testing

   * Aortic aneurysm >6cm
   * Unstable cardiovascular disease (unstable angina, myocardial infarction or pulmonary embolism <4 weeks prior)
   * Severe aortic stenosis
   * Pneumothorax
   * Cerebral aneurysm
   * Thoracic or abdominal surgery <4 weeks prior
4. Contra-indications to passing oesophageal balloons

   * Oesophageal ulceration or varices
   * Sinusitis, recent nasal surgery or epistaxis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects over the age of 16 with either chronic airflow obstruction or COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2021-08-22 (Estimated); Study Completion 2022-02-02 (Estimated)

PRIMARY OUTCOMES:
Respiratory resistance at 5Hz - 20Hz (R5-R20) (kPa/l/s) related to airtrapping as determined by quantitative CT (Expiratory phase low attenuation area <856 HU (%LAA <856 HU) | Baseline, pre-procedure
  Impulse Oscillometry

SECONDARY OUTCOMES:
Respiratory reactance at 5Hz: X5 (kPa/l/s) | Baseline, pre-procedure
  Impulse Oscillometry
Reactance area: Ax (kPa/l/s) | Baseline, pre-procedure
  Impulse Oscillometry
Functional residual capacity by MBNW: FRCgas (L) | Baseline, pre-procedure
  Multiple Breath Nitrogen Washout
Lung clearance index: LCI | Baseline, pre-procedure
  Multiple Breath Nitrogen Washout
Ventilation heterogeneity conducting airways: Scond (L/s) | Baseline, pre-procedure
  Multiple Breath Nitrogen Washout
Ventilation heterogeneity acinar airways: Sacin (L/s) | Baseline, pre-procedure
  Multiple Breath Nitrogen Washout
Forced expiratory volume in 1 second: FEV1 (L) | Baseline, pre-procedure
  Spirometry
Forced vital capacity: FVC (L) | Baseline, pre-procedure
  Spirometry
Total lung capacity: TLC (L) | Baseline, pre-procedure
  Plethysmography
Residual volume: RV (L) | Baseline, pre-procedure
  Plethysmography
Functional residual capacity by plethysmography: FRCpleth (L) | Baseline, pre-procedure
  plethysmography
Airway mean luminal diameter (Dmean) | Baseline, during the procedure
  Optical Coherence Tomography
Airway inner lumen area (Ai) | Baseline, during the procedure
  Optical Coherence Tomography
Airway wall area (Aw), airway wall percentage (Aw%) as determined by [Aw/(Ai + Aw) × 100%] | Baseline, during the procedure
  Optical Coherence Tomography
Air trapping - expiratory phase low attenuation area <856 HU (%LAA <856 HU) | Baseline, pre-procedure
  Quantitative CT
Modified MRC dyspnoea score | Baseline, pre-procedure
  Patient reported outcome measure
St George's Respiratory Questionnaire Score | Baseline, pre-procedure
  Patient reported outcome measure
Asthma-related Quality of Life Questionnaire (AQLQ) (if asthmatic) | Baseline, pre-procedure
  Patient reported outcome measure
Asthma Control Questionnaire (ACQ) (if asthmatic) | Baseline, pre-procedure
  Patient reported outcome measure
6-minute walk distance (m) | Baseline, pre-procedure
  6-minute walk distance (m)

OTHER OUTCOMES:
Exploratory: Inflammatory and pathological studies of airways brush, wash and cryobiopsy samples | Baseline, during the procedure
  Laboratory based scientific studies

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Brompton, London, United Kingdom